CLINICAL TRIAL: NCT01261624
Title: A Multicenter, Open Label, Dose Finding Study to Evaluate Efficacy and Safety of Givinostat Administered in Two Different Doses in Patients With Poly JIA Not Adequately Responding to the Standard Treatment.
Brief Title: Efficacy and Safety Dose Finding Study of Givinostat to Treat Polyarticular Course Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary reason for the decision to discontinue the study is lack of enrolment; this decision is not related to any tolerability concerns with Givinostat
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSC/08/2357/36
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Polyarticular Course Juvenile Idiopathic Arthritis
Keywords: poly JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Givinostat 1.0 mg/kg daily (Experimental)
  Interventions: Drug: Givinostat
- Givinostat 1.5 mg/kg daily (Experimental)
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — 1.0 mg/kg daily (0.5 mg/kg twice a day) in fed condition 1.5 mg/kg daily (0.75 mg/kg twice a day) in fed condition

SUMMARY:
The present study has been designed in order to evaluate the efficacy and safety of two doses of Givinostat in subjects with polyarticular course JIA

Givinostat ready-to-use suspension especially intended for paediatric administration, will be administered orally at different daily doses.

Patients with an established diagnosis of one of the following JIA forms (Polyarticular JIA rheumatoid factor positive or negative, Oligoarticular extended JIA, Systemic JIA without active systemic features) will be enrolled.

The treatment regimen will remain unchanged for 12 weeks and the clinical response will by assessed by applying the ACR Pediatric response criteria. Patients achieving at least an ACR Pediatric 30 response will continue receiving the assigned dose for 12 further weeks.

After the end of study (week 24) responder patients will be allowed to extend the treatment until they maintain a clinical benefit.

DETAILED DESCRIPTION:
Non-clinical data on Givinostat, support a potent anti-inflammatory mechanism of action which can potentially slow the arthritic destructive process. This rationale seems to be confirmed by the preliminary evidences collected in a previous Phase II clinical trial conducted in children and young adults with systemic JIA.

The present protocol is aimed at collecting new information on safety and efficacy of two doses of Givinostat for the treatment of JIA.

ELIGIBILITY:
Inclusion Criteria:

* patients of both genders, aged 2 to 17 years, with established diagnosis of polyarticular course Juvenile Idiopathic Arthritis (see before for specific subtypes) according to ILAR (International League Against Rheumatism) criteria (Petty RE et al., 2004) for at least six months before the study entry
* age at polyarticular JIA diagnosis < 16 years
* active disease for at least 6 months prior to enrolment as defined by the following criteria:
* presence of at least 5 active joints (those with swelling or, in the absence of swelling, limited range of motion accompanied by pain/tenderness)
* inadequate response to, or intolerance to, at least one biologic agent such as, but not limited to, etanercept, inﬂiximab, and adalimumab.
* maximum allowed steroid dose 0.2 mg/kg/day or 10 mg/day (whichever is lower) of prednisone or equivalent
* in case of concomitant methotrexate treatment, it has to be on a stable dose ≤15 mg/m2 weekly for at least 1 month before patient's enrolment
* other disease-modifying anti-rheumatic drugs possibly previously introduced have to be discontinued for a period of at least five half-lives
* concomitant nonsteroidal anti-inflammatory drugs, if any, on a stable dose for at least four weeks before patient's enrolment

Exclusion Criteria:

* patient with fever related to JIA or other systemic features of JIA during 12 months before entering the study
* active bacterial or mycotic infection requiring antimicrobial treatment
* episode of macrophage activation syndrome in the last 6 months
* a baseline prolongation of QT/QTc interval, use of concomitant medications that prolong the QT/QTc interval or history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) (Appendix C)
* clinically significant cardiovascular disease
* clinically significant illness i.e. any condition (including laboratory abnormalities) that in the opinion of the Investigator places the patient to unacceptable risk for adverse outcome if he/she were to participate in the study
* psychiatric illness/social situations that would limit compliance with study medication and protocol requirements
* inherited metabolic diseases
* presence of malignancy
* pregnancy or lactation
* positive blood test for HIV
* active EBV infection, active B and/or C hepatitis
* platelet count <100x109/L
* absolute neutrophil count <1.5x109/L
* serum creatinine >2xULN (Upper limit of normal).
* total serum bilirubin >1.5xULN.
* serum AST/ALT > 3xULN.
* congenital heart and/or central nervous system disorders

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zulian, MD, Principal Investigator — Azienda Ospedaliera-Università di Padova - Unità di Reumatologia Pediatrica
Locations (13):
- Universitair Ziekenhuis Gent, Ghent, Gent, Belgium
- 1st Faculty of Medicine and General Faculty Hospital, Prague, Prague, Czechia
- Italy (4):
  - Ospedale Meyer, Florence, FI
  - Policlinico G. Martino, Messina, ME
  - Istituto Gaetano Pini, Milan, MI
  - Azienda Ospedaliera-Università di Padova, Padua, PD
- Romania (2):
  - Institutul pentru Ocrotirea Mamei si Copilului "Alfred Rusescu", Bucharest, București
  - Spitalul Clinic de Urgenta pentru Copii "M.S. Curie", Bucharest, București
- Serbia (3):
  - Institute of Rheumatology Belgrade, Belgrade, Belgrade
  - Mother and Child Health Institute "Dr Vukan Cupic", New Belgrade, Belgrade
  - University Clinical Center Nis, Niš, Nis
- Children's Hospital - University Medical Centre Ljubljana, Ljubljana, Ljubljana, Slovenia
- Hospital Ramón y Cajal, Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2010 - December 2011. The study was conducted by nine Investigators in five countries across Europe; three Investigators in Italy, two Investigators each in Romania and Serbia, and one Investigator each in Czech Republic and Slovenia
Groups:
- Low Dose Treatment Cohort (LDTC): 0.50 mg/kg Twice Daily (BID): Patients (pts) received the dose of 0.50 mg/kg BID for 12 weeks in fed condition
- High Dose Treatment Cohort (HDTC): 0.75 mg/kg BID: Patients received the dose of 0.75 mg/kg BID for 12 weeks in fed conditions
Period: Week 0 to Week 12
Arm/Group | Low Dose Treatment Cohort (LDTC): 0.50 mg/kg Twice Daily (BID) | High Dose Treatment Cohort (HDTC): 0.75 mg/kg BID
Started | 10 | 6
Completed | 9 | 3
Not Completed | 1 | 3
Not completed — Disease Progression | 1 | 1
Not completed — Insufficient Response | 0 | 2
Period: Week 13 to Week 24
Arm/Group | Low Dose Treatment Cohort (LDTC): 0.50 mg/kg Twice Daily (BID) | High Dose Treatment Cohort (HDTC): 0.75 mg/kg BID
Started | 1 (Of 9 pts from LDTC: 5 non-responders switched to HDTC; 4 pts responded, but 3 switched to HDTC) | 11 (Of 6 pts of HDTC: 3 non-responders went out of study, 3 continued. 8 swithched from LDTC to HDTC)
Completed | 1 | 10
Not Completed | 0 | 1
Not completed — Insufficient Response | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Treatment Cohort (LDTC): 0.50 mg/kg BID: Patient received the dose of 0.50 mg/kg for 12 weeks in fed condition
- High Dose Treatment Cohort (HDTC): 0.75 mg/kg BID: Patient received the dose of 0.75 mg/kg for 12 weeks in fed condition
- Total: Total of all reporting groups
Arm/Group | Low Dose Treatment Cohort (LDTC): 0.50 mg/kg BID | High Dose Treatment Cohort (HDTC): 0.75 mg/kg BID | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (5.5) | 9.7 (5.7) | 10.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Serbia | 5 | 1 | 6
  Czech Republic | 1 | 1 | 2
  Slovenia | 1 | 1 | 2
  Romania | 1 | 0 | 1
  Italy | 2 | 3 | 5
Body Weight [Mean (Standard Deviation); unit: kg] | 37.36 (15.40) | 37.92 (18.59) | 37.57 (16.05)
Height [Mean (Standard Deviation); unit: m] | 1.388 (0.204) | 1.365 (0.277) | 1.379 (0.225)

OUTCOME MEASURES:

1. Primary Outcome: ACR Pediatric Response Level (ACRPRL) 30 After 12 Weeks of Treatment
Description: ACR Pediatric variables include: Physician's Global Assessment of disease activity on a 0-100 mm visual analogue scale from 0 mm = no disease activity to 100 mm = very severe disease activity; Parent's or patient's Global Assessment of Patient's overall well-being on a 100 mm VAS from 0 mm = very well to 100 mm = very poor; Functional ability: Childhood Health Assessment Questionnaire; Number of joints with active arthritis using the ACR definition (any joint with swelling, or in the absence of swelling, limitation of motion accompanied by pain/tenderness not due to bone deformity); Number of joints with limitation of motion; Laboratory measure of inflammation: C-reactive protein (mg/L) Patients were considered as responders if they achieve at least an ACR Pediatric Criteria level 30 of response, defined as a 30% improvement as compared to baseline in at least 3 of the 6 variables listed above, with no more than 1 variable worsening by > than 30%
Time Frame: 12 weeks of treatment
Measure: Number; unit: participants
Groups:
- Low Dose Discontinued: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Of the 10 pts enrolled to initial Low Dose treatment cohort (LD), 1 pt discontinued the study before wk 12 (Low Dose Discontinued treatment cohort).
- Low Dose Throughout: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Of the 10 patients enrolled to initial Low Dose treatment cohort 4 pts achieved ACR Pediatric Criteria level 30 of response at Week 12, one of them continued the same dose for further 12 weeks (Low Dose Throughout treatment cohort)
- Switched Dose: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Of the 10 patients enrolled to initial Low Dose treatment cohort, 4 pts achieved ACR Pediatric Criteria level 30 of response at Week 12, 3 of them switched to the high dose at the Investigator's decision for further 12 weeks agreed by the Sponsor (Switched Dose treatment cohort).
- High Dose Throughout: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Six patients were enrolled to initial High Dose treatment cohort; two patients continued the same dose throughout the study (High Dose Throughout treatment cohort)
- High Dose Discontinued: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Six patients were enrolled to initial High Dose treatment cohort; four patients discontinued the study (High Dose Discontinued treatment cohort
Arm/Group | Low Dose Discontinued | Low Dose Throughout | Switched Dose | High Dose Throughout | High Dose Discontinued
Number analyzed (Participants) | 1 | 1 | 8 | 2 | 4
participants
  ACR Pediatric Response Level 30 | 0 | 1 | 3 | 2 | 1
  No response | 1 | 0 | 5 | 0 | 3

2. Secondary Outcome: ACR Pediatric Response Level (ACR 50, 70, 90 and 100) at Week 12
Description: ACR Pediatric variables include: Physician's Global Assessment of disease activity on a 0- 100 mm visual analogue scale from 0 mm = no disease activity to 100 mm = very severe disease activity; Parent's or patient's Global Assessment of Patient's overall well-being on a 100 mm VAS from 0 mm = very well to 100 mm = very poor; Functional ability: Childhood Health Assessment Questionnaire; Number of joints with active arthritis using the ACR definition (any joint with swelling, or in the absence of swelling, limitation of motion accompanied by pain/tenderness not due to bone deformity); Number of joints with limitation of motion; Laboratory measure of inflammation: C-reactive protein (mg/L) Patients were considered as responders if they achieve at least an ACR Pediatric Criteria level 50, 70, 90 and 100 of response, defined as a 50%, 70%, 90% and 100% improvement as compared to baseline in at least 3 of the 6 variables listed above, with no more than 1 variable worsening by > than 30%
Time Frame: at week12
Measure: Number; unit: participants
Arm/Group | Low Dose Discontinued | Low Dose Throughout | Switched Dose | High Dose Throughout | High Dose Discontinued
Number analyzed (Participants) | 1 | 1 | 8 | 2 | 4
participants
  ACR Pediatric response Level 50 | 0 | 1 | 1 | 2 | 1
  ACR Pediatric response Level 70 | 0 | 1 | 0 | 1 | 0
  ACR Pediatric response Level 90 | 0 | 0 | 0 | 0 | 0
  ACR Pediatric response Level 100 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Planned treatment duration was 24 weeks overall (12 weeks + 12 weeks). The mean (SD) duration of treatment was 131.9 (55.9) days overall, with a median duration of 170 days.
Description: All 16 pts experienced TEAEs; a total of 71 events: 5 (31.3%) pts experienced a total of 7 TEAEs considered related to the IMP. The severe TEAE experienced by 1 (6.3%) pt led to study discontinuation. No serious TEAEs or TEAEs with fatal outcome were reported.
Groups:
- Switched Dose: The initial two treatment cohorts were expanded in to 5 treatment cohorts for better evaluation of efficacy and safety end points. Of the 10 patients enrolled to initial Low Dose treatment cohort, 4 pts achieved ACR Pediatric Criteria level 30 of response at Week 12, 3 of them switched to the high dose at the Investigator's decision for further 12 weeks agreed by the Sponsor (Switched Dose treatment cohort). Safety data selected for high and low dose in this cohort are not available, this kind of analysis has not been performed.
Arm/Group | Low Dose Discontinued | Low Dose Throughout | Switched Dose | High Dose Throughout | High Dose Discontinued
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/8 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 8/8 | 2/2 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Discontinued (N=1) | Low Dose Throughout (N=1) | Switched Dose (N=8) | High Dose Throughout (N=2) | High Dose Discontinued (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coxsackie Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation Irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less